CLINICAL TRIAL: NCT00863785
Title: Treatment of Acute Severe Alcoholic Hepatitis With Corticoids Plus N Acetyl Cysteine Versus Corticoids Alone: a French Multicentre Randomized Controlled Study.
Brief Title: Treatment of Severe Alcoholic Hepatitis With Corticoids Plus N Acetyl Cysteine Versus Corticoids Alone
Acronym: HAA-NAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Amiens University Hospital, Amiens University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHRC R04 - Dr NGUYEN-KHAC; AFSSAPS 040276
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: Alcoholic Hepatitis
Keywords: Acute Alcoholic Hepatitis; Cirrhosis; Alcohol; Alcoholic Liver disease
MeSH Terms: conditions — Hepatitis, Alcoholic; Fibrosis; Liver Diseases, Alcoholic | interventions — Adrenal Cortex Hormones; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Corticoids plus N Acetyl Cysteine (Experimental): 40 mg/d prednisolone N Acetyl Cysteine infusion 150mg/kg in 30 minutes then 50 mg/kg in 4 h then 100mg/kg in 16 h and finally 100mg/d2 to d5
  Interventions: Drug: Corticoids plus N Acetyl Cysteine

INTERVENTIONS:
Drug: Corticoids plus N Acetyl Cysteine — 40 mg/d prednisolone N Acetyl Cysteine infusion 150mg/kg in 30 minutes then 50 mg/kg in 4 h then 100mg/kg in 16 h and finally 100mg/d2 to d5
  Other Names: AAH-NAC study

SUMMARY:
35% of Acute Alcoholic Hepatitis patients (AAH) do not respond to corticoids and died after 6 months. Chronic alcohol abuse depletes glutathione in the hepatocytes and makes the latter more sensitive to excessive TNFα levels. Re-establishment of a stock of antioxidants by administration of a precursor (N-acetyl cysteine, NAC) in combination with corticoids (C) could make the hepatocytes more resistant and improve survival. The investigators' study's primary endpoint was improvement of survival at 6 months. The secondary endpoints were survival at 1 and 3 months, tolerance of NAC and a drop in blood bilirubin levels at D7

DETAILED DESCRIPTION:
AAH patients (Maddrey score > 32 and compatible histological results) should centrally randomized into the C-NAC or C groups. Both groups received 4 weeks of prednisolone treatment, plus NAC for the combination therapy group (D1: 150, 50 and 100 mg/kg in 250, 500 and 1000 mL of 5% glucose-saline (G5%) respectively, at t=30 minutes, 4 and 16 hours; D2 to D5, 100 mg/kg in 1000 mL of G5%). Group C received 1000 mL of G5%, D1-5

ELIGIBILITY:
Inclusion Criteria:

* Patient consent
* Chronic alcohol intake in the last 3 to 6 months
* Maddrey score ≥ 32
* Liver histology compatible

Exclusion Criteria:

* Hepato renal syndrome
* Hepatocarcinoma
* Recent variceal haemorrhage
* Recent bacterial infections
* Other liver diseases associated (HCV, HBV, hemochromatosis, AIH)
* Cancers or cardiac and respiratory, HIV infection
* NAC Allergy
* No patient consent
* Acetaminophen intoxication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2004-04; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Survival at one, three and six months | six months

SECONDARY OUTCOMES:
bilirubin decrease at day seven survival at one and three months nac tolerance side effects | one, three and six months

CONTACTS AND LOCATIONS:
Overall Officials: Phillippe DOMY, Study Director — Centre Hospitalier Universitaire, Amiens
Locations (13):
- France (13):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Centre Hospitalier Beauvais, Beauvais
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire de Caen, Caen
  - Centre Hospitalier de Cambrai, Cambrai
  - Centre Hospitalier de Compiègne, Compiègne
  - Centre Hospitalier de Lens, Lens
  - Centre Hospitalier Saint-Antoine, Paris
  - Centre Hospitalier Universitaire Pitié-Salpétrière, Paris
  - Centre Hospitalier Universitaire de Reims, Reims
  - Centre Hospitalier Universitaire de Rouen, Rouen
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
  - Centre Hospitalier de Valenciennes, Valenciennes

REFERENCES:
- [Derived] Nguyen-Khac E, Thevenot T, Piquet MA, Benferhat S, Goria O, Chatelain D, Tramier B, Dewaele F, Ghrib S, Rudler M, Carbonell N, Tossou H, Bental A, Bernard-Chabert B, Dupas JL; AAH-NAC Study Group. Glucocorticoids plus N-acetylcysteine in severe alcoholic hepatitis. N Engl J Med. 2011 Nov 10;365(19):1781-9. doi: 10.1056/NEJMoa1101214. PMID 22070475